CLINICAL TRIAL: NCT01137201
Title: Internal Hernia After Laparoscopic Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Erik Stenberg, MD, MD, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPN 2009/415
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: The Prevalence of Surgery for Small Bowel Obstruction After LGBP Procedure.
Keywords: Small bowel obstruction; Laparoscopic gastric bypass; Internal Hernia; Mesenteric defect; Morbid obesity
MeSH Terms: conditions — Internal Hernia; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenteric defects sutured (Experimental): Closure of the mesenteric defects using running, non-absorbable suture
  Interventions: Procedure: Suturing of mesenteric defects
- Mesenteric defects not sutured (No Intervention): Non-closure of the mesenteric defects

INTERVENTIONS:
Procedure: Suturing of mesenteric defects
  Arms: Mesenteric defects sutured

SUMMARY:
To see if closing the mesenteric defects created at a Laparoscopic Gastric Bypass is better than leaving them open.

DETAILED DESCRIPTION:
When the patients who has undergone a Laparoscopic Gastric Bypass lose weight, the mesenteric defects that are inevitable to cause, gets bigger and can cause an internal hernia (IH). This study will observe whether it is better to close the defects or leave them open. The patients will be randomized into two groups. One, where the defects are closed with sutures and one where the defects are left alone. The primary endpoint of the study is the prevalence of surgery for obstruction. Information about this will be gathered through the national register for obesity surgery in Sweden, SOReg. Each arm in the study will include 1200 patients and the follow up period will be three years. Since the register mentioned above is an ongoing register, the results can be studied over a longer period if wanted. The national hospital registry will further improve the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Any patient accepted for a Laparoscopic Gastric Bypass that has given a written consent

Exclusion Criteria:

* Conversion to open surgery prior to the randomization
* Patients not giving a written consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2507 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Surgery for small bowel obstruction after a LGBP procedure. | 2 years

SECONDARY OUTCOMES:
Serious Complications | within 2 years after surgery
  Defined as Clavien grade 3b or more

CONTACTS AND LOCATIONS:
Overall Officials: Ingmar Näslund, MD, PhD, Study Director — Scandinavian Obesity Surgery Registry
Locations (1):
- Department of Surgery, Örebro University Hospital, Örebro, Örebro County, Sweden

REFERENCES:
- [Derived] Stenberg E, Ottosson J, Magnuson A, Szabo E, Wallen S, Naslund E, Thorell A, Naslund I. Long-term Safety and Efficacy of Closure of Mesenteric Defects in Laparoscopic Gastric Bypass Surgery: A Randomized Clinical Trial. JAMA Surg. 2023 Jul 1;158(7):709-717. doi: 10.1001/jamasurg.2023.1042. PMID 37163240
- [Derived] Stenberg E, Szabo E, Ottosson J, Thorell A, Naslund I. Health-Related Quality-of-Life after Laparoscopic Gastric Bypass Surgery with or Without Closure of the Mesenteric Defects: a Post-hoc Analysis of Data from a Randomized Clinical Trial. Obes Surg. 2018 Jan;28(1):31-36. doi: 10.1007/s11695-017-2798-z. PMID 28676957
- [Derived] Stenberg E, Szabo E, Agren G, Ottosson J, Marsk R, Lonroth H, Boman L, Magnuson A, Thorell A, Naslund I. Closure of mesenteric defects in laparoscopic gastric bypass: a multicentre, randomised, parallel, open-label trial. Lancet. 2016 Apr 2;387(10026):1397-1404. doi: 10.1016/S0140-6736(15)01126-5. Epub 2016 Feb 16. PMID 26895675